CLINICAL TRIAL: NCT07170072
Title: Community-based Evaluation of a Novel, System-wide Harm Reduction Strategic Plan for People Experiencing Homelessness in New York City
Brief Title: Shelter HArm Reduction Evaluation
Acronym: SHARE
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 24-01708; R01CE003699 (NIH)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Overdose; Harm Reduction
MeSH Terms: conditions — Drug Overdose; Harm Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Aims 1a, 1b, and 2: Individuals in the NYC Single-Adult Homeless Services: Investigators will conduct an analysis of administrative data on the population of individuals in the NYC single-adult homeless services system during 2021-2026.
- Aim 3: Homeless Services Clients Staff: Qualitative interviews and focus group sessions will be held with homeless services providers and administrators who have delivered the HRSP interventions.
- Aim 3: Homeless Services Clients: Qualitative interviews and focus group sessions will be held with homeless clients who have received one or more of the HRSP interventions.
- Aim 3: Homeless Services Stakeholders: Qualitative interviews and focus group sessions will be held with stakeholders, who work in a role in which they have key insight to the HRSP interventions, including planning and implementation.

SUMMARY:
The proposed study will use mixed methods research to examine overdose and other health-related impacts of harm reduction initiatives in NYC homeless shelters.

DETAILED DESCRIPTION:
Mixed-methods study using analyses of administrative homeless services and Medicaid data (Aims 1a, 1b, and 2) and in-depth qualitative interviews (Aim 3). This study will examine the implementation and impact of a Harm Reduction Strategic Plan (HRSP) portfolio of interventions in the NYC single-adult shelter system. The study will be conducted using administrative data (Aims 1a, 1b, and 2) and in-depth interviews and focus groups about client and staff experiences with the HRSP.

ELIGIBILITY:
Inclusion Criteria:

For Aims 1a, 1b, and 2: There will be no participant enrollment or direct contact with individuals as these aims will involve the use of an analytic dataset comprised of linked administrative NYC homeless services, Medicaid, and vital records. The dataset will include records for individuals who entered the NYC DHS single-adult shelter system during calendar years 2021-2026, as well as a matched comparison group(s) (as identified through Medicaid data) during the same years. The matched comparison group will be comprised of individuals age 18 and older with active Medicaid coverage at the time of observation.

For Aim 3 Homeless Services Client participant group: To be eligible for participation in this study, an individual must meet all of the following criteria:

* Adult 18 year of age or older
* Speak English
* Is staying or has stayed in an NYC single-adult shelter that has implemented HRSP interventions
* Report past-year drug use
* Able and willing to provide consent

For Aim 3 Homeless Services Staff participant group: To be eligible for participation in this study, an individual must meet all of the following criteria:

* 18 years of age or older
* Speak English
* Works at an adult shelter service provider agency that implemented HRSP or received HRSP interventions (role may include case manager, security staff, shelter director, medical staff, organizational leadership)
* Able and willing to provide consent

For Aim 3 Homeless Services Stakeholder participant group: To be eligible for participation in this study, an individual must meet all of the following criteria:

* 18 years of age or older
* Speak English
* Works in a role in which they have key insight to the HRSP interventions, including planning and implementation (role may include homeless services administrator or other key stakeholder)
* Able and willing to provide consent

Exclusion Criteria:

Aims 1a, 1b, and 2: Children under age 18 years of age will be excluded.

Aim 3: Under age 18 years old, currently a prisoner (we are not sampling from locations where we expect to encounter prisoners), unable to communicate in English (because the interview and focus group guides will not be validated for use in other languages), and unable to provide informed consent.

For Aim 3 Homeless Services Client participant group: those who are not staying or have not stayed at a shelter with HRSP interventions and those who do not report past-year drug use will not be excluded.

For Aim 3 Homeless Services Staff participant group: those who have not been employed in a shelter with the HRSP interventions will be excluded. In alignment with standard techniques of purposeful sampling and the study goal of ensuring a range of experiences is captured in the qualitative interviews, additional targeting or exclusion criteria might be set by investigators as needed to ensure that a diverse range of experiences is included among qualitative interview participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aims 1a, 1b, and 2: Analysis of administrative data will include the population of individuals in the NYC single-adult homeless services system during 2021-2026.
  Aim 3: Qualitative interview and focus group participants will include homeless clients who have received one or more of the HRSP interventions and homeless services providers and administrators who have delivered the HRSP interventions.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Fatal Overdose (OD) | Day 0 (Administrative Analysis of Data)
Incidence of Non-Fatal Overdose (OD) | Day 0 (Administrative Analysis of Data)

SECONDARY OUTCOMES:
Incidence of Substance Use Disorder (SUD) Treatment Initiation | Day 0 (Administrative Analysis of Data)
Incidence of Health Services Utilization | Day 0 (Administrative Analysis of Data)

CONTACTS AND LOCATIONS:
Overall Officials: Bennett Allen, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This study is not a clinical trial and is not subject to data sharing requirements. The study involves qualitative interviews with sensitive information and data will not be shared outside of the research team in line with confidentiality agreements and restrictions outlined in our IRB approval.